CLINICAL TRIAL: NCT02192476
Title: Efficacy of California Tri-pull Taping Method in the Treatment of Post Stroke Shoulder Subluxation- A Randomized Clinical Trial.
Brief Title: Efficacy of CTPT Method in the Treatment of Post Stroke Shoulder Subluxation
Acronym: CTPT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Subhasish Chatterjee, SUBHASISH CHATTERJEE, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTPT
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Subluxation of Inferior Shoulder
Keywords: Stroke, subluxation
MeSH Terms: conditions — Stroke; Joint Dislocations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional (Active Comparator): 15 participants are allotted in this arm and each participants received conventional neuro rehabilitation programme 5 days a week for 6 weeks.
  Interventions: Other: conventional neuro rehabilitation programme
- intervention (Experimental): 15 participants allotted in this arm and each participants received California tri-pull taping method along with conventional neuro rehabilitation was given 5 days a week for 6 weeks
  Interventions: Other: conventional neuro rehabilitation programme; Other: California tri-pull taping (CTPT)

INTERVENTIONS:
Other: conventional neuro rehabilitation programme — All the conventional group subjects were received standardized conventional neuro rehabilitation programme. The conventional neuro rehabilitation treatment includes, active, and passive range of motion exercise, bilateral activation of pectoralis major, activation of latissimus dorsa, activation of the retractors, weight bearing exercise of upper extremity, activation of supraspinatus, reaching activities, grasping, holding and release, and activity of daily living (ADL) activities. Every participant was received conventional neuro rehabilitation for 45 minutes and 5 days a week.
Other: California tri-pull taping (CTPT) — Two types of tape was used, a self-adhesive 1.5" cotton undercover tape and a 1" rigid strapping tape. Participants placed their affected arm on a supporting surface to better approximate the humeral head back into the glenoid fossa. The three pieces of rigid tape were applied to the patient's shoulder on top of the already applied self-adhesive cotton tape.
  Arms: intervention

SUMMARY:
california tri-pull taping (CTPT) method might be effective in reducing shoulder subluxation, pain, and improving active flexion range (AFLXN) range of motion, and functional recovery after stroke.

DETAILED DESCRIPTION:
All the experimental group participants will receive conventional neuro rehabilitation for 45 minutes along with California tri-pull taping on the subluxed extremity. Lead researcher applied the CTPT method. The tape was applied as following manner.

Before the first intervention day, participants with hair on their shoulder or upper arm were asked to shave the area. Two types of tape was used, a self-adhesive 1.5" cotton undercover tape and a 1" rigid strapping tape. Participants placed their affected arm on a supporting surface to better approximate the humeral head back into the glenoid fossa. The three pieces of rigid tape were applied to the patient's shoulder on top of the already applied self-adhesive cotton tape. The first piece (medial) was applied from 1.5" below the deltoid tuberosity running straight up the middle of the arm to 2" above the top of the glenoid fossa between the clavicle and the spine of the scapula. The second piece (posterior) was located from 1.5" below the deltoid tuberosity to 1.5" above the middle of the spine of the scapula. The medial border of this second piece ran along the acromial process. Last, the third piece (anterior) was located from 1.5" below the deltoid tuberosity to run around the front of the humeral head and over the coracoid process, up to 1.5" above the clavicle. The tape will removed and new tape applied every Monday, Wednesday, and Friday and remained on the patient for 6 consecutive weeks.

Following the 6 weeks, each patients of both group was individually re-assessed and evaluated the effect of intervention and parameters were recorded. The recording and measurement obtained before and after intervention was subjected to statistical analysis and the result of that interpreted to obtain the significance of study.

ELIGIBILITY:
Inclusion Criteria:

1. Acute stroke.
2. A minimum of 5 mm (0.2 in) shoulder subluxation in the involved upper extremity.
3. Mini mental status examination (MMSE) score >23.
4. Age (35-70 yrs.) and of either sex.
5. Brunnstroms stage 1 and 2. -

Exclusion Criteria:

1. Mini mental status examination (MMSE) score <23.
2. Other musculoskeletal disorder of the affected upper extremity.
3. History of trauma to the affected upper extremity.
4. Hyper or hypo sensitivity disorders.
5. Any skin allergy.
6. Brunnstorm's stage 3 and 4.
7. Individual affected from neurological disorder other than stroke.
8. Un-cooperative patients.
9. Individuals with psychosomatic disorder

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Digital Vernier caliper. | 6 month
  Digital Vernier caliper (Aerospace super) is used to measure the accromion- humeral distance in shoulder subluxation patients.

SECONDARY OUTCOMES:
Universal Goniometer | 6 month
  Universal Goniometer is used to measure the active shoulder flexion range of motion (AFLXN). The measurement is taken in lying position.
Fugl-Meyer scale (FUG) | 6 month
  FUG scale was used to measure the upper extremity motor recovery.
Visual analogue scale (VAS) | 6 month
  VAS was used to measure the post stroke shoulder subluxation pain.

CONTACTS AND LOCATIONS:
Overall Officials: Senthil P Kumar, PhD, Study Director — MMIPR
Locations (1):
- MMIPR, Ambāla, Haryana, India